CLINICAL TRIAL: NCT03854331
Title: OBEAT - Beating Obesity: A Feasibility Trial
Brief Title: OBEAT - Beating Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: TRYG Foundation (Other); Oak Foundation (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Berit Lilienthal Heitmann, Professor, Principal investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TRYG-125690
Record Dates: First submitted 2019-02-04; First posted 2019-02-26 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy Related; Obesity, Childhood; Stress
Keywords: Resilience; Cortisol; Feasibility; Healthy lifestyle; Sleep
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resilience program (Experimental): The resilience program consists of different modules that are based on research on mentalization, mindfulness, parent management training, improving self-control and self-efficacy, cognitive behaviour therapy, social learning theory and neuroscience. The MyResilience program is also informed by cognitive bias modification and self-control training research. These techniques have been found to be effective in improving engagement in health behaviours and reducing symptoms and negative behaviours in clinical groups
  Interventions: Behavioral: Resilience program
- Standard care (No Intervention): Danish antenatal standard care is 3 visits at the general practitioner, 5 midwife controls and 2 ultrasound scans

INTERVENTIONS:
Behavioral: Resilience program — The resilience program consists of different modules that are based on research on mentalization, mindfulness, parent management training, improving self-control and self-efficacy, cognitive behaviour therapy, social learning theory and neuroscience. The MyResilience program is also informed by cognitive bias modification and self-control training research. These techniques have been found to be effective in improving engagement in health behaviours and reducing symptoms and negative behaviours in clinical groups
  Arms: Resilience program

SUMMARY:
The primary objective of this trial is to study the feasibility of a resilience intervention to reduce stress and thus improve sleep, healthy diet and physical activity in normal weight pregnant women.

Initially, an exploratory study of stressors and worrying in pregnant women will be done by use of qualitative methods (focus group interviews) followed by a randomised controlled feasibility trial with a parallel qualitative process evaluation.

This project is expected to improve the understanding of the processes and feasibility of conducting a randomized intervention study to examine if improvements in chronic stress and poor sleep during pregnancy improves early weight gain and childhood risk of obesity.

DETAILED DESCRIPTION:
Phase 1: Planning In Phase 1 (6 months), the project will be developed and planned, and approvals from the Danish Data Protection Agency and Ethical Committee of the Capital Region to conduct the study will be obtained.

Validated questionnaires to measure perceived stress, sleep patterns, physical activity- and dietary habits will be selected and pilot tested.

Phase 2: Recruitment and data collection In Phase 2 (12 months), participants will be recruited and randomized. Pregnant women living in Denmark are offered public, antenatal care delivered by hospital employed midwives. Healthy, non-obese, pregnant women assigned to antenatal care and birth at Hvidovre Hospital, are routinely invited to a first antenatal midwife session at gestational week 14-18. At these sessions, participants will be informed and recruited to the feasibility study. In 8 weeks approximately 240 pregnant women will be eligible, thus 120 women corresponding to 50% of all eligible pregnant women in one month will be recruited. In this feasibility study 50% of the women will be randomised to the intervention group and introduced to the resilience internet-based program/ smart phone app and 50% will be randomised to the control group and receive standard care. Computer-based randomization procedures will be used.

Phase 3: Feasibility study evaluation In Phase 3 (19 months), the knowledge obtained in Phase 2 will be evaluated.

An effect evaluation of the project will be conducted by analysing the collected clinical data, primarily related to changes and correlations in chronic stress in mother and infant (measured by hair cortisol), perceived stress, physical activity- and dietary habits, infant birth length and weight, and gestational age.

A process evaluation will also be conducted. The Committee of Health Education will collect data on how much and what parts of the resilience program has been used by the participating pregnant women. In addition, the participants will be asked to complete a short questionnaire on how frequent and how satisfied they have been with using the program. The researchers also want to use qualitative focus group interviews to investigate the participants' attitudes and acceptability of the proposed intervention.

The results of the effect- and process evaluations will be synthesized and will, depending on the results of the feasibility study, be implemented in a following planning of a large RCT.

Qualitative analytical methods The interview guide will be developed based on a literature search of existing literature in the field. To minimize the bias of my own influence I will consider my own experience and pre-understanding as a midwife.

The interviews will be recorded digitally and subsequently transcribed literally. The data will be analyzed using content analysis as described by Graneheim & Lundman. The purpose of the content analysis is to organize and understand the meaning of the data collected in the focus group interviews and to draw conclusions from it.

Statistical analysis The clinical outcomes will be examined using paired t-tests as well as linear or logistic regression analyses. Analyses will be done crude and adjusted for potential confounders obtained from the completed questionnaires. Results of the analyses of the clinical outcomes are expected to be underpowered due to the feasibility design of this study but will however provide estimates indicating any direction or effect size of the resilience program on this target group.

ELIGIBILITY:
Inclusion Criteria:

* Expecting first child
* Speaks Danish
* Non-obese (BMI < 30)
* Singleton pregnancy
* Visited to basic level midwife care

Exclusion Criteria:

* Non-danish speakers
* Type 1 or 2 diabetes
* Visited to specialist midwife care for psychosocial reasons
* Expecting twins
* BMI > 30
* Multipara

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Recruitment-rates - feasibility | Two months after birth
  Number of participants out of eligible pregnant women approached
Recruitment-time - feasibility | Two months after birth
  Number of days used to recruit the decided number of 120 participants
Attrition-rates - feasibility | Two months after birth
  Number of participants leaving the study before the end
Follow up-rates - feasibility | Two months after birth
  Number of participants in final clinical examination
Compliance-rates - feasibility | Two months after birth
  Use of resilience program measured from web-statistics
Self-reported compliance-rates - feasibility | Two months after birth
  Use of resilience program from patient-reported questionnaire
Satisfaction-rates - feasibility | Two months after birth
  Measured from patient-reported questionnaire

SECONDARY OUTCOMES:
Change in maternal chronic stress | Gestational week 14-18, 28, 35, birth and two months after birth
  Assessed by level of cortisol (ng/ml) in 3 cm scalp hair
Change in maternal perceived stress | Gestational week 14-18, 28, 35 and two months after birth
  Assessed by Cohen's Perceived Stress Scale (PSS). PSS measures the respondent's experience of stress over the past four weeks using ten questions to answer to what extent the respondent experiences his life as unpredictable, uncontrollable and stressful, and whether he or she feels nervous or stressed. The scale goes from 0 to 40. The higher the score, the higher the level of stress experienced.
Change in maternal depression, anxiety and tension/stress. | Gestational week 14-18, 28, 35 and two months after birth
  Assessed by The Depression and Anxiety Stress Scale (DASS). DASS is a 42-item self report instrument designed to measure the three related negative emotional states of depression, anxiety and tension/stress. The scale goes from 0 to 42 for every emotional state. The higher the score, the higher the level of depression, anxiety or stress experienced. Range: Stress: Normal 0-10, Mild 11-18, Moderate 19-26, Severe 27-34, Extremely severe 35-42.
  Anxiety: Normal 0-6, Mild 7-9, Moderate 10-14, Severe 15-19, Extremely severe 20-42.
  Depression: Normal 0-9, Mild 10-12, Moderate 13-20, Severe 21-27, Extremely severe 28-42.
Change in mentalization ability | Gestational week 14-18, 28, 35 and two months after birth
  Assessed by the Reflective Functioning Questionnaire, which comprises eight items and includes two subscales: Certainty (RFQc) and uncertainty (RFQu) about mental states. The 7 point Likert scale contains answers ranging from strongly disagree to strongly agree. Of the 6 items on each subscale, two are unique and four shared across the two scales. With the RFQc subscale, strong disagreement reflects hypermentalizing, and agreement to any degree (or a neutral response) reflects more genuine mentalizing (acknowledging the opaqueness of mental states). With the RFQu subscale, high agreement scores reflect a stance characterised by a lack of knowledge about mental states, or 'hypo-mentalizing', and lower scores represent an acknowledgement of the opaqueness of mental states, a characteristic of good mentalizing. Both scales are based on a mean of the 6 items (Cucchi et al. (2018), PeerJ, DOI 10.7717/peerj.5756).
Changes in maternal Sense of Coherence (SOC) | Gestational week 14-18, 28, 35 and two months after birth
  Assessed by Antonovsky's 13-item SOC scale, which measures comprehensibility (5 items), manageability (4 items), and meaningfulness (4 items). Each item has seven graded (Likert-type) response scale, which is summed up and the total scores can range from 13 (low SOC) to the maximum of 91 (highest possible SOC).
Changes in maternal resilience | Gestational week 14-18, 28, 35 and two months after birth
  Assessed by the Connor-Davidson Resilience Scale (CD-risc). The scale comprises of 25 items, each rated on a 5-point scale (0-4). The total score ranges from 0-100, with higher scores reflecting greater resilience.
Differences in parental stress | Two months after birth
  Assessed by The Parental Stress Scale (PSS). PSS is made up of 18 items rated on a Likert- type 5-point scale that describes the parent-child relationship and how each parent feels about it. A higher score indicates a higher level of parental stress.
Changes in fear of childbirth | Gestational week 14-18, 28, 35
  Fear of childbirth is assessed asking the question 'Are you anxious about the course of the upcoming delivery?' in a participant-reported questionnaire. Possible responses are: 'Not at all', 'A little' or 'A lot'. Only the last response is considered to represent fear of childbirth.
Changes in fetal health anxiety | Gestational week 14-18, 28, 35
  Fetal health anxiety is assessed asking the question 'Are you anxious about the health of the expected child?' in a participant-reported questionnaire. Possible responses are: 'Not at all', 'A little' or 'A lot'. Only the last response is considered to represent fetal health anxiety.
Sleep patterns - mother | Gestational week 14-18, 28, 35 and two months after birth
  Self-reported sleep duration and sleep quality measured from participant-reported questionnaire
Changes in participant's physical activity - transportation | Gestational week 14-18, 28, 35 and two months after birth
  Self-reported means of transportation (biking, public transportation, car, walking) in hours pr. week
Changes in participant's physical activity - exercise | Gestational week 14-18, 28, 35 and two months after birth
  Self-reported exercise (i.e. dancing, yoga or badminton) in hours pr. week
Changes in diet - mother | Gestational week 14-18, 28, 35 and two months after birth
  Measured with a Food Frequency Questionnaire (FFQ) developed for the Danish National Birth cohort is used for dietary assessment. Most questions focus on the dietary habits during the 4 weeks prior to completion of the questionnaire, but a number of questions address changes in dietary habits during pregnancy. The FFQ includes questions on intake of 360 food and beverage items in the previous 4 weeks and is validated with a 7-day weighted food record. The 360 food items recorded in the FFQ are aggregated into 36 food groups and, together with the daily intake (in grams) for each food group, eaten by a given individual, are used to identify dietary patterns.
Weight - mother | Gestational week 14-18, 28, 35 and two months after birth
  Maternal weight (kg) measured at midwife sessions
Weight - child | Birth and two months after birth
  Weight (kg), obtained from birth records and clinical examination
Length - child | Birth and two months after birth
  Length (cm) obtained from birth records and clinical examination
Head circumference - child | Birth and two months after birth
  Head circumference (cm) obtained from birth records and clinical examination

OTHER OUTCOMES:
Diet - infant (breastfeeding, bottlefeeding) | Two months after birth
  Measured from participant-reported questionnaire
Infant crying | Two months after birth
  Measured from participant-reported questionnaire in hours of crying pr. day
Differences in infant chronic stress | Birth and two months after birth
  Level of cortisol (ng/ml) in 3 cm scalp hair
Differences in birth method | Birth
  Vaginal birth, elective cesarean og acute cesarean obtained from birth records
Differences in epidural-rate | Birth
  Epidural as pain relief during birth from birth records
Differences in rates of prolonged labour | Birth
  Use of oxytocin-drip during birth from birth records
Differences in use of private healthcare providers | Gestational week 14-18, 28, 35, birth and two months after birth
  Yes/no in participant-reported questionnaire
Differences in absence from work during pregnancy | Gestational week 14-18, 28, 35
  Reasons to absence (i.e. pregnancy complications) and number of days absent in participant-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Berit Heitmann, Professor, Principal Investigator — Research Unit for Dietary Studies at The Parker Institute Bispebjerg and Frederiksberg Hospital
Locations (1):
- Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ladekarl M, Specht IO, Adegboye ARA, Brodsgaard A, Nohr EA, Olsen NJ, Heitmann BL. The feasibility of a web-based resilience-building program to prevent stress among danish pregnant nulliparous women: A randomised controlled feasibility trial. PLOS Ment Health. 2025 Sep 8;2(9):e0000294. doi: 10.1371/journal.pmen.0000294. eCollection 2025. PMID 41661987
- [Derived] Ladekarl M, Olsen NJ, Winckler K, Brodsgaard A, Nohr EA, Heitmann BL, Specht IO. Early Postpartum Stress, Anxiety, Depression, and Resilience Development among Danish First-Time Mothers before and during First-Wave COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Nov 9;18(22):11734. doi: 10.3390/ijerph182211734. PMID 34831493